CLINICAL TRIAL: NCT03557788
Title: Changes in Microbiota and Metabolomic Profile Between Rifaximin Responders and Non-responders In Diarrhoea-Predominant Irritable Bowel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017/00977
Record Dates: First submitted 2018-05-02; First posted 2018-06-15 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: Rifaximin
MeSH Terms: interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rifaximin (Experimental): Patients who receive PO Rifaximin 500mg TDS for 2 weeks. All patients will receive treatment to evaluate the effect of the intervention. This is a single-arm study.
  Interventions: Drug: Rifaximin Oral Tablet

INTERVENTIONS:
Drug: Rifaximin Oral Tablet — PO 550mg TDS for 2 weeks

SUMMARY:
Irritable Bowel Syndrome (IBS) carries a high prevalence worldwide and imposes substantial economic burden on patients, healthcare systems and society. In recent years, dysbiosis of the gut microbiota and bile acid (BA) malabsorption have been identified as putative pathophysiological mechanisms. Bile acid metabolism and gut microbiota are closely related. When patients with IBS-D were compared to healthy subjects, total levels of faecal BAs do not differ, but increased faecal primary BAs and reduced secondary BAs have been repeatedly observed in patients with IBS-D, suggesting abnormal BA deconjugation. Rifaximin, a non-absorbable antibiotic, has been shown in a recent meta-analysis to produce a therapeutic clinical gain compared to other treatment options for IBS, including placebo, paralleled by a high safety profile. It is also now known that changes in fecal microbiota have been observed in patients with IBS who have responded positively to Rifaximin. The relationship between microbiota changes, metabolomics changes after Rifaximin is unclear. There is emerging data to suggest duodenal dysbiosis as a putative pathophysiology, which in one study, clustered together with salivary microbiota than with fecal microbiota. However, the oral microbiome in patients with IBS has never been explored, which could possibly explain the downstream observations of duodenal and fecal dysbiosis. The investigators aim to assess the changes in metabolomic and microbiota profile after Rifaximin treatment, between responders and non-responders. The investigators will also explore the oral microbiome in IBS patients, and assess its relationship with fecal microbiome between responders and non-responders.

DETAILED DESCRIPTION:
The primary hypothesis of the study is that amongst responders to Rifaximin, fecal primary BAs will be significantly reduced, and faecal secondary BAs significantly increased after treatment.

The secondary hypotheses include:

1. Reduction in Escherichia and increase in Lactobacillus after treatment, as a possible mechanism to explain the increased deconjugation of primary BAs observed.
2. Oral microbiome correlates with gut microbiome dysbiosis in IBS-D subjects.
3. Rifaximin therapy alters both oral and gut microbiota, and that responders to Rifaximin harbour different microbiota compared to non-responders.

   1. Primary Objectives Primary Objective: To compare oral microbiome and fecal microbiome in IBS-D patients before and after Rifaximin, examining differences between responders and non-responders.
   2. Secondary Objectives Secondary objectives: To examine the differences between stool and salivary metabolomics, urinary metabolomics and serum immunomics and metabolomics, between responders and non-responders to Rifaximin in IBS-D subjects.

Responders to Rifaximin will be defined as patients having a 50 point or more reduction in the IBS Symptom Severity Score (IBS-SSS) after treatment. This indicates that the patient has experienced a significant improvement in the reduction of symptoms. The IBS-SSS is a well-validated questionnaire that is patient-administered. This questionnaire will be administered at Day 0 and Day 14 of Rifaximin.

Up to 50 subjects with Diarrhoea-predominant Irritable Bowel Syndrome (IBS-D) will be recruited from the National University Hospital Gastroenterology clinic and Singapore General Hospital Gastroenterology clinic. There will be subject restrictions on race, so as to limit variation due to inter-racial differences and ensure homogeneity in the subject population.

Determination of Sample Size Adopted from the sample size calculation table for human microbiome studies by La Rosa (La Rosa et al. 2012), the study will require 15 subjects to have 80% power at p<0.05 significance level. To account for multiple testing, investigators will require at least 25 subjects for each category to have 90% power at p<0.01 significance level. The investigating team will be recruiting a total of 40 respondents and 40 non-respondents from both NUH and SGH.

Statistical and Analytical Plans Pair-wise comparison will be conducted between the 2 sample groups for differences in the microbiome. Concordance will be examined between the oral and fecal groups, both before and after treatment. Identified species will be examined for possible metabolic pathways based on their genetic profiles generated by the metagenomic analysis.

Data Quality Assurance Demographics will be collected from the patient medical records. The oral conditions will be recorded in data collection form after oral examinations. The data collection form will be checked and signed off by PI. All the records will be entered twice into database by the delegated study team members to ensure accuracy of data.

Data Entry and Storage Initial collection will be on paper-based data collection form. All subjects will be assigned a unique study subject code and the data collection form will be labelled with subject recruitment number. The de-identified data will be transferred into analysis software and kept on an encrypted flash drive kept by the delegated study team members. The data collection form will be put in lockable cabinet for 6 years after study completion, being accessed by study team only. De-identified data may be provided to a biostatistician for further analysis.

Study Visits and Procedures This is a multi-centre open-label prospective cohort study. Recruited subjects will be patients who are newly diagnosed IBS-D, who undergo a two-week course of Rifaximin as indicated by their primary physician. Patients with symptomatic improvement (responders) after treatment will be compared to patients who do not improve (non-responders), based on a validated IBS Symptom Severity Score. As this is a cohort study, there will be no randomization or blinding. All patients will receive Rifaximin and no placebo will be used.

The study will consist of the following phases:

Visit 1: Screening The screening phase will include assessing eligibility based on the inclusion and exclusion criteria, obtaining informed consent, followed by a one-week symptom, bowel and 3-day dietary diary. All subjects will undergo further oral examination to determine oral status such as caries and periodontal status. This is to accurately evaluate the patient's baseline symptoms, bowel and dietary habits. Patients will be given a stool collection kit for collection of stool sample (10-20g) to be returned before or at the next visit.

Visit 2: Enrolment and treatment (Day 1 Rifaximin) After the screening phase, patients will complete the IBS-SSS, and will be enrolled if a score of 300 or greater is obtained. Urine (50ml), saliva (5-10ml), 2 buccal swabs and blood samples (20ml) will be obtained during this visit as well.

Patients will then initiate Rifaximin for two weeks. During these two weeks, patients will continue the symptom, bowel and 3-day dietary dairy, and also whether they have remembered to take their medication, and any side effects observed.

Visit 3: Follow-up post-treatment (Day 14 Rifaximin) Patients will be asked to provide stool (10-20g), urine (50ml), saliva (5-10ml), 2 buccal swabs and blood samples (20ml) again at or 1-week after Day 14, and repeat the IBS-SSS. The diaries will be collected, and compliance to medication will be verified.

Subjects who discontinue the study early due to an AE will be followed until resolution or stabilization of the event.

Visit 4: Review of symptoms 90 days after completing Rifaximin treatment. Patients will be asked to repeat the IBS-SSS. The symptom, bowel and 3-day dietary dairy will be collected and patients will be asked to provide stool (10-20g), urine (50ml), saliva (5-10ml), 2 buccal swabs and blood samples (20ml).

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study if he/she meets all of the following criteria:

  1. Chinese subjects between 21 to 65 years of age.
  2. Male or female Females of childbearing (reproductive) potential must have a negative serum pregnancy test at screening and agree to use an acceptable method of contraception throughout their participation in the study. Acceptable methods of contraception include double barrier methods (condom with spermicide jelly or diaphragm with spermicide), hormonal methods (oral contraceptives, patches or medroxyprogesterone acetate), or an intrauterine device (IUD) with a documented failure rate of less than 1% per year. Abstinence may be considered an acceptable method of contraception at the discretion of the investigator.

     Note: Females who have been surgically sterilized (eg, hysterectomy or bilateral tubal ligation) or who are postmenopausal (total cessation of menses for >1 year) will not be considered "females of childbearing potential".
  3. Subject has IBS-D confirmed by the Rome III or IV diagnostic criteria below:

     a. Rome IV Criteria: i. Recurrent abdominal pain, on average, at least 1 day per week in the last 3 months, associated with 2 or more of the following criteria:

  <!-- -->

  1. Related to defecation
  2. Associated with a change in frequency of stool
  3. Associated with a change in form (appearance) of stool ii. Criteria fulfilled for the last 3 months with symptom onset at least 6 months before diagnosis b. Rome III Criteria: i. Recurrent abdominal pain or discomfort at least 3 days/month in the last 3 months associated with two or more of the following:

  <!-- -->

  1. Improvement with defecation
  2. Onset associated with a change in frequency of stool
  3. Onset associated with a change in form (appearance) of stool ii. Criterion fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis iii. "Discomfort" means an uncomfortable sensation not described as pain. iv. Pain/discomfort frequency of at least 2 days a week. c. IBS-Diarrhoea (IBS-D) i. Predominant bowel habits are based on stool form on days with at least one abnormal bowel movement. Subtyping based on at least 2 weeks of daily diary data is recommended, using the "25% rule." Subtyping established when the patient is evaluated off medications used to treat bowel habit abnormalities. Patients must have more than 25% of bowel movements with Bristol stool form types 6 or 7 and less than 25% of bowel movements with Bristol stool form types 1 or 2.
  4. Subject does not have adequate relief of IBS symptoms on the first day of screening (Day 0) and has an IBS-SSS of at least 300 out of 500.
  5. Subject had a colonic evaluation (either colonoscopy or CT Colonography) within the last 5 years as part of an evaluation for IBS or IBS symptoms (which excludes inflammatory or neoplastic disease).
  6. Subject must maintain a stable diet for the duration of the study.
  7. Subject is capable of understanding the requirements of the study, is willing to comply with all study procedures, understands the language of the informed consent form, and is capable and willing to sign the informed consent form.

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if he/she meets any of the following criteria:

  1. Subject has other forms of IBS (Constipation predominant, Alternating, or Mixed)
  2. Subject has failed to record at least 3 days of the daily diary assessments during the Screening Phase.
  3. Subject has current evidence of duodenal ulcer, gastric ulcer, diverticulitis, or infectious gastroenteritis. Note: Subjects with gastroesophageal reflux disease controlled by stable doses of medication or diet are eligible to participate in the study
  4. Subject has a history of inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis, celiac disease), GI malignancy, GI obstruction, gastroparesis, carcinoid syndrome, pancreatitis, amyloidosis, ileus or cholelithiasis
  5. Subject has diabetes (Type 1 or Type 2)
  6. History of surgery to remove a segment of the gastrointestinal tract or bariatric surgery for obesity, or cholecystectomy at any time
  7. Appendectomy within 2 months or other abdominal surgeries within 6 months before entry into the trial
  8. Subject has a positive stool test for Yersinia enterocolitica, Campylobacter jejuni, Salmonella, Shigella, ovum and parasites, and/or Clostridium difficile
  9. Subject who has psychiatric disorders which are not controlled ("controlled" is based on the Investigator's medical judgment); subjects with psychoses are excluded regardless of current therapy.
  10. Subject has current or recent history (within 12 months before signing informed consent) of drug, laxative or alcohol abuse
  11. Subject is pregnant or lactating
  12. Subject has a history of human immunodeficiency virus (HIV) or hepatitis (B or C)
  13. Subject has a history of abnormal thyroid function not controlled by thyroid medications
  14. Subject has unstable cardiovascular or pulmonary disease, categorized by a worsening in the disease condition that required a change in treatment or medical care within 1 month of randomization
  15. Subject has known allergy to rifaximin or rifampin or excipients
  16. Subject has participated in an investigational drug or device study within the 30 days prior to signing informed consent
  17. Subject has active malignancy within the last 5 years (exceptions: basal cell carcinomas of the skin, or if female, in situ cervical carcinoma that has been surgically excised)
  18. Subject has ever taken Rifaximin prior to this study
  19. Antibiotics and probiotic consumption within the last1 month.
  20. Drugs that could alter GI transit time or microbiome, or bile acid sequestrants. These include antidiarrheals (eg, loperamide), narcotics, prokinetic drugs.

NOTE: Tricyclic antidepressants and serotonin re-uptake inhibitors are allowed if the subject is at stable doses for at least 6 weeks prior to signing informed consent and the dose will remain stable throughout the duration of the study.

Medication to be avoided

The following concomitant medications are to be avoided if possible, after initiation of the diary eligibility period and throughout the study:

* Any experimental drugs
* Probiotic supplements
* Antibiotics
* Antipsychotic drugs
* Antispasmodics
* Antidiarrheals (eg, loperamide and bismuth subsalicylate)
* IBS drugs (e.g., Alosetron)
* Lubiprostone
* Narcotics (specifically opioid analgesics)
* Prokinetic drugs
* Warfarin
* Nonsteroidal anti-inflammatory drugs are prohibited if used for the treatment of IBS

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in IBS-SSS questionnaire | Start of Rifaximin treatment (Visit 2, which is 1 week after first/screening visit), End of Rifaximin treatment (Visit 3, which is 2 weeks after Visit 2), and 3 months after end of treatment (Visit 4)
  Severity of IBS-D will be measured using IBS-SSS questionnaire, at baseline (visit 2) and at completion of 2 week course of Rifaximin (Visit 3) as well as 3 months after end of Rifaximin (Visit 4). A responder will be defined as a reduction of IBS-SSS by more than 50 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Soh Yu Sen, Alex, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No